CLINICAL TRIAL: NCT00006063
Title: Randomized Study of Pancrelipase With Bicarbonate (PANCRECARB) Capsules in Reducing Steatorrhea in Patients With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Indiana University School of Medicine (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15154; IUMC-9506-10; DIGEST-97-0001-1B
Record Dates: First submitted 2000-07-05; First posted 2000-07-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-07

CONDITIONS: Cystic Fibrosis
Keywords: cardiovascular and respiratory diseases; cystic fibrosis; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases | interventions — Pancrelipase; Bicarbonates

INTERVENTIONS:
Drug: pancrelipase with bicarbonate

SUMMARY:
OBJECTIVES:

I. Compare the efficacy of enteric coated pancrelipase with bicarbonate (PANCRECARB) capsules versus the patient's usual enteric coated pancreatic enzyme without bicarbonate in decreasing fecal fat and nitrogen losses in patients with cystic fibrosis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, multicenter study. In the first treatment period, patients are randomized to one of two treatment arms.

Arm I: Patients receive enteric coated pancrelipase with bicarbonate (PANCRECARB) capsules before meals and snacks for 7 consecutive days.

Arm II: Patients receive their usual enteric coated pancreatic enzyme without bicarbonate capsule before meals and snacks for 7 consecutive days.

Patients receive approximately 50% of their usual lipase dose during treatment. Food intake is recorded on days 1-3, food intake is weighed and recorded on days 4-7, and stools are collected over 72 hours on days 5-7 to determine fecal fat and nitrogen excretion. Anthropometric measurements including height, weight, and skinfolds are assessed.

In the second treatment period, patients are switched to the alternate treatment arm after a 3 day washout period. Patients receive the opposing treatment as per protocol.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Clinical diagnosis of cystic fibrosis Duplicate sweat chloride measurements greater than 60 mEq/L on samples collected after pilocarpine iontophoresis
* Patients with a history of malabsorption who consume at least 1,000 to 2,500 lipase units/kg/meal

--Prior/Concurrent Therapy--

* No concurrent oral antibiotics, antacids, H2 receptor antagonists, or any drugs known to interfere with digestion

--Patient Characteristics--

* Weight for height greater than the 5th percentile
* No prior meconium ileus with intestinal resection
* No known hypersensitivity to pancrelipase or pork protein

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Start 1999-07; Study Completion 1999-08

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sue Brady, Study Chair — Indiana University School of Medicine